CLINICAL TRIAL: NCT02019641
Title: The NIH Exercise Therapy for Advanced Lung Disease Trials: Response and Adaptation to Aerobic Exercise in Patients With Interstitial Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Inova Fairfax Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 140027; 14-CC-0027
Record Dates: First submitted 2013-12-20; First posted 2013-12-24 (Estimated); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2022-06

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Interstitial Pneumonitis; Desquamative Interstitial Pneumonia
Keywords: Exercise; Interstitial Lung Disease; Pulmonary Rehabilitation
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Interstitial Pneumonitis, Desquamative, Familial; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Intervention (AET+) (Experimental): Participant with interstitial lung disease performed aerobic exercise three times a week plus weekly education for 10 weeks
  Interventions: Other: Aerobic Exercise Training (AET); Other: Education
- Control Group (CON) (Active Comparator): Participant with interstitial lung disease performed weekly education for 10 weeks, then crossed over to perform aerobic exercise three times a week for 10 weeks
  Interventions: Other: Education

INTERVENTIONS:
Other: Aerobic Exercise Training (AET) — walking on a treadmill at vigorous intensity for up to 45 minutes
  Arms: Aerobic Exercise Intervention (AET+)
Other: Education — Weekly education

SUMMARY:
Interstitial lung disease (ILD) is the result of over 200 etiological pathways arising from several different insults to the lung parenchyma: inhaled substances, drug side effects, connective tissue disease, infection, and malignancy. The disease can also be of idiopathic origin. If prolonged, the resulting inflammation causes permanent and progressive fibrotic reorganization of the parenchyma and small airways, which reduces the distensibility of the lung and impedes O2 and carbon dioxide (CO2) exchange.

This study is a randomized controlled trial to determine the safety and efficacy of aerobic exercise for patients who have interstitial lung disease (ILD) uncomplicated by pulmonary hypertension. In an uncontrolled study, we observed more efficient cardiorespiratory function, increased physical work capacity, and improved health-related quality of life following aerobic exercise in this study population. Serious adverse events resulting from aerobic exercise training were not observed and our work to date has established plausibility for the efficacy of aerobic exercise training and its safety for patients with ILD.

DETAILED DESCRIPTION:
There are two primary treatment conditions. Patients with ILD are be randomized to either an intervention consisting of aerobic exercise training plus patient education or a control condition that includes patient education only. Aerobic exercise training will consist of a 10-week regimen of supervised treadmill walking three times a week. The duration of the exercise sessions will progress from 30 minutes to 45 minutes per session over the 10 weeks, as tolerated. The intensity of the exercise will be determined based on results of a cardiopulmonary exercise test. Those randomized to control will not initially engage in aerobic exercise training. There will, however, be a secondary study: a crossover design in which subjects in the control group will complete the aerobic exercise regimen.

* Participants must be between the ages of 21 and 80 and live within a reasonable travel distance from the greater Washington D.C. area
* All pre and post testing will be conducted at the NIH Clinical Center in Bethesda, Maryland. Each testing session will last about 6 hours and will consist of a medical history and examination; six questionnaires on health, fatigue, activity, and mood; electrocardiogram, transthoracic echocardiogram, pulmonary function tests, six-minute walk test (6MWT); and urine pregnancy test (if applicable). Other required tests are:
* A maximum treadmill test: The exercise begins at an easy level and gradually increases until the participant says he or she can no longer continue or the investigator decides it is not safe to continue. Participants are fitted with a mask, electrodes and light sensors to measure how well the heart is working and how well the muscles use oxygen.
* An arterial occlusion muscle oxygenation capacity test:: During seated rest, a light sensor that measures the oxygen level in the muscle is placed on the calf while a pressure cuff will then be placed around the thigh. The cuff is rapidly inflated and held at a high pressure for up to 10 minutes and then deflated.
* A blood sample for complete blood count and Nt-ProBNP (a hormone that indicates damage to heart muscle).
* Aerobic exercise training and education may take place at either the NIH Clinical Center in Bethesda, Maryland, or the Pulmonary Rehabilitation Program at INOVA Fairfax Hospital in Falls Church, Virginia.

ELIGIBILITY:
* INCLUSION CRITERIA:

A diagnosis of interstitial lung disease, including idiopathic pulmonary fibrosis (IPF), non-specific interstitial pneumonitis (NSIP), sarcoidosis, or other form of chronic lung fibrosis based on clinical context via clinic note from a pulmonologist.

Individuals with ILD referred for pulmonary rehabilitation who are 21-80 years of age and live in the Washington metropolitan area.

No episodes of fainting or significant chest pain for at least one month.

No prior pulmonary rehabilitation received within the last 6 months and not currently in a maintenance program.

Physically inactive (no participation in a structured exercise program as defined as more than 30 minutes of exercise 3 or more days a week within the last 6 months).

EXCLUSION CRITERIA:

Other medical conditions that would impair aerobic capacity or the ability to engage in physical activity, including other pulmonary, cardiovascular, neurological, musculoskeletal or metabolic conditions

Other medical conditions that may pose a risk to exercise testing or training as determined by the investigators (for example, peripheral vascular disease)

Diagnosis of pulmonary hypertension

Inability to maintain a resting oxygen saturation greater than or equal to 90% SpO2, measured by pulse oximetry on supplemental oxygen

Inability to complete a treadmill cardiopulmonary exercise test.

Significant hepatic or renal dysfunction.

Metastatic cancer with a life expectancy of less than one year.

Active substance abuse.

Severe psychiatric disease

Antiretroviral therapy

Pregnancy

Ongoing tobacco use

Acceptance onto a lung transplant waiting list

Active participation in ILD drug trials

Inability to read English

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-05-23 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - INOVA Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified scientific data (e.g., 6 minute-walk test distance, clinical tests, survey questionnaires) will be made available at the discretion of the Principle Investigator.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available when the resources become available to perform the deidentification. The data will available until Jan. 1st, 2028.
Access Criteria: De-identified scientific data may be shared directly with those requesting it as deemed appropriate by the Principle Investigator on a resource available basis.

REFERENCES:
- [Background] Chan L, Chin LMK, Kennedy M, Woolstenhulme JG, Nathan SD, Weinstein AA, Connors G, Weir NA, Drinkard B, Lamberti J, Keyser RE. Benefits of intensive treadmill exercise training on cardiorespiratory function and quality of life in patients with pulmonary hypertension. Chest. 2013 Feb 1;143(2):333-343. doi: 10.1378/chest.12-0993. PMID 22922554
- [Background] Keyser RE, Woolstenhulme JG, Chin LM, Nathan SD, Weir NA, Connors G, Drinkard B, Lamberti J, Chan L. Cardiorespiratory function before and after aerobic exercise training in patients with interstitial lung disease. J Cardiopulm Rehabil Prev. 2015 Jan-Feb;35(1):47-55. doi: 10.1097/HCR.0000000000000083. PMID 25313451
- [Background] Keyser RE, Christensen EJ, Chin LM, Woolstenhulme JG, Drinkard B, Quinn A, Connors G, Weir NA, Nathan SD, Chan LE. Changes in fatigability following intense aerobic exercise training in patients with interstitial lung disease. Respir Med. 2015 Apr;109(4):517-25. doi: 10.1016/j.rmed.2015.01.021. Epub 2015 Feb 7. PMID 25698651
- [Background] Weinstein AA, Chin LM, Keyser RE, Kennedy M, Nathan SD, Woolstenhulme JG, Connors G, Chan L. Effect of aerobic exercise training on fatigue and physical activity in patients with pulmonary arterial hypertension. Respir Med. 2013 May;107(5):778-84. doi: 10.1016/j.rmed.2013.02.006. Epub 2013 Mar 7. PMID 23478192
- [Background] Morris ZV, Chin LMK, Chan L, Guccione AA, Ahmad A, Keyser RE. Cardiopulmonary exercise test indices of respiratory buffering before and after aerobic exercise training in women with pulmonary hypertension: Differentiation by magnitudes of change in six-minute walk test performance. Respir Med. 2020 Apr;164:105900. doi: 10.1016/j.rmed.2020.105900. Epub 2020 Feb 25. PMID 32217288
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-CC-0027.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 46 subjects consented, 11 subjects met exclusion and one self-withdrew prior to randomization.
Groups:
- Control Group (CON) Then AET: Participant with interstitial lung disease that crossed over from the control arm to perform aerobic exercise three times a week for 10 weeks
Period: 10-Week Follow up
Arm/Group | Aerobic Exercise Intervention (AET+) | Control Group (CON) | Control Group (CON) Then AET
Started | 17 | 17 | 0
Completed | 14 | 16 | 0
Not Completed | 3 | 1 | 0
Not completed — Withdrawal by investigator | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Period: 20-Week Follow up
Arm/Group | Aerobic Exercise Intervention (AET+) | Control Group (CON) | Control Group (CON) Then AET
Started | 0 | 0 | 15
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by investigator | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise Intervention (AET+) | Control Group (CON) | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 9 | 10 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 9 | 8 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-minute Walk Test Distance (6MWD)
Description: The 6-minute walk test (6MWT) is a measure of physical capacity and subjects are instructed to walk as far as possible around a pre-measured walking course over a time period of six minutes. The 6-minute walk test distance (6MWD) is the total distance walked in meters during the 6MWT and greater distance walked means better physical capacity. This outcome is reported as the difference between time-points (post- minus pre-10 weeks).
Time Frame: Before and after 10 weeks
Population: The analyses included only those subjects who completed the 6MWT at both time points (baseline and after 10-weeks)
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Aerobic Exercise Intervention (AET+) | Control Group (CON)
Number analyzed (Participants) | 14 | 16
Meters | 46.5 (35.8) | 23.2 (38.6)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Aerobic Exercise Intervention (AET+) | Control Group (CON) | Control Group (CON) Then AET
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 1/15
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/17 | 2/15
Other Adverse Events (participants affected / at risk) | 1/17 | 0/17 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Intervention (AET+) (N=17) | Control Group (CON) (N=17) | Control Group (CON) Then AET (N=15)
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Intervention (AET+) (N=17) | Control Group (CON) (N=17) | Control Group (CON) Then AET (N=15)
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated early due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT02019641/Prot_SAP_000.pdf